CLINICAL TRIAL: NCT06118645
Title: An Open, Multicenter, Phase II Study of Cadonilimab Combined With Paclitaxel (Albumin-bound) in the Treatment of Advanced Gastric Adenocarcinoma or Esophagogastric Junction Adenocarcinoma With PD-(L)1 Inhibitors Resistance
Brief Title: Cadonilimab+ Paclitaxel (Albumin-bound) Treat Advanced Gastric Adenocarcinoma With PD-(L)1 Inhibitors Resistance
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jingdong Zhang, Clinical Professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-025
Record Dates: First submitted 2023-09-10; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gastric Adenocarcinoma
Keywords: cadonilimab; paclitaxel (albumin-bound); gastric adenocarcinoma; PD-(L)1 inhibitors resistance; esophagogastric junction adenocarcinoma

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open, multicenter clinical study to evaluate the efficacy and safety of cadonilimab in combination with paclitaxel (albumin-bound type) as a second-line treatment for advanced gastric adenocarcinoma or esophagogastric junction adenocarcinoma The study included a screening period (no more than 28 days after the subject signed the informed consent letter to the first dose) treatment period (receiving the appropriate treatment regimen until the disease progression and toxicity of intolerable withdrawal of the informed consent letter and death or the end of the study, whichever occurred first) and follow-up period (including safety follow-up and survival follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadonilimab combined +paclitaxel (albumin-bound) (Experimental): cadonilimab combined +paclitaxel (albumin-bound)
  Interventions: Drug: cadonilimab combined +paclitaxel (albumin-bound)

INTERVENTIONS:
Drug: cadonilimab combined +paclitaxel (albumin-bound) — 1. In the safe induction phase6 subjects will receive cadonilimab (10mg/kg, Q3W, intravenous infusion, up to 2 years) and paclitaxel (albumin-bound type)(125 mg/m2,Days1, 8,Q3w, intravenous infusion, up to 8 cycles).
  2. If the safety and tolerability are good, and the initial efficacy signal is observed, the extended enrollment phase will enter the extended enrollment phase of drug administration and the safety introduction phase

SUMMARY:
Cadonilimab combined with paclitaxel (albumin-bound) treat advanced gastric adenocarcinoma or esophagogastric junction adenocarcinoma with PD-(L)1 inhibitors resistance

DETAILED DESCRIPTION:
An open, multicenter, Phase II study of cadonilimab combined with paclitaxel (albumin-bound) in the treatment of advanced gastric adenocarcinoma or esophagogastric junction adenocarcinoma that has failed prior treatment with PD-(L)1 inhibitors

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign a written informed consent, which must be signed prior to performing the specified study procedure required for the study.
2. Age and gender: ≥18 years old and≤75 years old, both men and women.
3. The Eastern United States Cancer Collaborative (ECOG) physical Fitness score was 0-1.
4. Histologically or cytologically confirmed unresectable or metastatic gastric adenocarcinoma or esophagogastric junction adenocarcinoma (EGJ defined as the center of the tumor within 5 cm of the anatomic location of the cardia, as described in the Siewert classification system).
5. Patients who have progressed or become intolerant after prior treatment with a regimen containing PD-1/PD-L1 monoclonal antibody had a tumor shrinkage response assessed as CR, PR, or reduced SD(<0% reduction in total target lesion diameter from baseline according to RECIST v 1.1) and persisted for 4 months or more after treatment with PD-1/PD-L1 monoclonal antibody If the disease progresses during neoadjuvant/adjuvant chemotherapy or radical chemoradiotherapy or within 6 months after the end of the last treatment, it is considered to have received first-line treatment
6. Expected survival ≥12 weeks.
7. According to RECIST v1.1, subjects must have at least one measurable lesion. For subjects who have previously received radiotherapy, a radiation-treated lesion may be considered a target if there is objective evidence of significant progression after radiotherapy if there is no other alternative target lesion.
8. Subjects are required to provide the most recent archived (at least 2 years old) and/or freshly obtained tumor tissue samples and at least 3 unstained FFPE pathological slides.
9. The functions of important organs must meet the following requirements:

(1) Hematological system: Neutrophil count≥1.5×10^9/L; Platelet count≥100×10^9/L; Hemoglobin≥90g/L; (2) Liver function： Serum albumin≥28g/L; Total bilirubin (TBI)≤1.5×ULN; Alanine aminotransferase (ALT)≤3×ULN (or≤5×ULN if liver metastates are present); Aspartate aminotransferase (AST)≤2.5×ULN (or≤5×ULN if liver metastates are present); (3) Renal function: Calculated creatinine clearance≥50 mL/min (using the Cockcroft-Gault formula); Female: CrCl = (140- age in years) × weight in kg × 0.85 72 × serum creatinine in mg/ dL

Male: CrCl = (140- age in years) × weight in kg × 1.00 72 × serum creatinine in mg/ dL

Urinary protein 2+ or 24 hours (h) urinary protein quantification<1.0g. (4) Coagulation function: Subjects not receiving anticoagulation therapy: INR or APTT ≤ 1.5×ULN; (5) Cardiac function: Left ventricular ejection fraction (LVEF)≥ 50 10. Fertile female subjects must undergo a urine or serum pregnancy test within 3 days prior to the first dosing (if the urine pregnancy test result is not confirmed negative, serum pregnancy test is required, based on the blood pregnancy result), and the result is negative if the fertile female subject is not neutered The subject must be on a highly effective contraceptive method since screening and must consent to continued use of the contraceptive method for 120 days after the last dose of the study drug; Whether to stop contraception after this time point should be discussed with the investigator.

11.If an unsterilized male subject has sex with a fertile female partner, the subject must use an effective contraceptive method from the beginning of screening until the 120th day after the last dose; Whether to stop contraception after this time point should be discussed with the investigator.

12.Subjects were willing and able to comply with the schedule for visiting treatment protocol laboratory tests and other study requirements.

Exclusion Criteria:

Patients with any of the following criteria were excluded from the study

1. Other pathological types confirmed by histopathological or cytological examination, such as squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma and Mixed pathological types will be judged according to the main components, adenocarcinoma components confirmed by the pathologist greater than 70% can be included in the group
2. Participants had other malignancies within 3 years prior to enrollment. Subjects with other malignancies that have been cured by local treatment, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical cancer, or carcinoma in situ of the breast, are not excluded.
3. The last systemic anti-tumor therapy, including chemotherapy and radiotherapy, immunotherapy, targeted therapy (small molecule targeted therapy is within 2 weeks before the first drug administration), and biologic therapy, was received within 3 weeks before the first drug administration; Palliative local treatment for non-target diseases and foci was performed within 2 weeks before the first administration; Received systemic non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, etc.) within 2 weeks prior to initial administration; Received Chinese herbal medicine or proprietary Chinese medicine with anti-tumor indications within 2 weeks prior to the first administration。
4. Previously received immunotherapy other than PD-1/PD-L1 inhibitors, including immune checkpoint inhibitors (such as anti-CTLA-4 antibodies, anti-CD47 antibodies, anti-SIRP-α antibodies, anti-LAG-3 antibodies, etc.), immune checkpoint agonists, and immune cell therapy Any treatment targeting the immune mechanism of tumor action.
5. Taxoids have been used in anti-tumor therapy in the past (including chemotherapy drugs such as paclitaxel and docetaxel)..
6. HER-2 overexpression (immunohistochemistry 2+ and FISH+, and immunohistochemistry 3+) did not use anti-HER-2 therapy (including trastuzumab, etc.) in previous anti-tumor therapy.
7. Any of the following has occurred during previous treatment with PD-1/PD-L1 inhibitors:

(1)There has been a history of grade 3 or higher irAE(excluding endosecretory system-related irAE) from PD-1/PD-L1 inhibitor therapy that resulted in permanent discontinuance of therapy, grade 2 immune-related cardiotoxicity, or any grade of neurological or ocular irAE; (2)Prior to screening in this study, subjects who were treated with prior PD-1/PD-L1 inhibitors and did not have complete remission of all adverse events or did not have remission to grade 1 were admitted to the study if their condition was stable and asymptomatic with appropriate alternative therapy; (3)Previous adverse events requiring immunosuppressant therapy other than glucocorticoids or recurrent adverse events during prior immunotherapy requiring systemic glucocorticoid therapy.

8. People with active autoimmune diseases that have required systemic treatment within the past two years (such as treatment with disease-modifying drugs, corticosteroids, immunosuppressive agents) and replacement therapy (such as thyroxine, islet, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered a systemic treatment.

9. Subjects with known active or untreated brain metastases, meningeal metastases, spinal cord compression, or pIA disease are admitted if they meet the following requirements and have measurable lesions outside the central nervous system: Asymptomatic after treatment, radiologically stable for at least 4 weeks prior to the start of study therapy (e.g. no new or enlarged brain metastases), and systemic glucocorticoid and anticonvulsant therapy have been discontinued for at least 2 weeks.

10. The presence of pleural effusion, pericardial effusion or peritoneal effusion with clinical symptoms requiring diuretic treatment and/or repeated drainage.

11. Clinically significant gastrointestinal obstruction, gastrointestinal perforation, intraperitoneal abscess, and fistula formation occurred within 6 months before first administration.

12. The presence of active or recurrent inflammatory gastrointestinal diseases (e.g. Crohn's disease ulcerative colitis radiation enteritis hemorrhagic enteritis chronic diarrhea, etc.) 13. History of myocarditis, cardiomyopathy, and malignant arrhythmias, Unstable angina pectoris requiring hospitalization, myocardial infarction, congestive heart failure (grade 2 or higher as defined by the New York Heart Association Functional Scale), or vascular disease (such as risk of rupture) in the 12 months prior to initial administration Aneurysms), or other heart damage that may affect the safety evaluation of the investigational drug (e.g., poorly controlled arrhythmias, myocardial ischemia).

14. Severe infection within 4 weeks prior to initial dosing, including but not limited to comorbiditic sepsis or severe pneumonia that requires hospitalization; Active infections that have received systemic anti-infective therapy within 2 weeks prior to initial dosing (excluding antiviral therapy for hepatitis B or C) 15. Subjects with known active tuberculosis (TB) and suspected active TB should be clinically screened for exclusion; Known active syphilis infection 16. Subjects with current active hepatitis B (HBsAg positive with more than 1000 copies /ml(200 IU/ml) of HBV-DNA or higher than the lower limit of detection, whichever is higher) are required to receive anti-HBV therapy during the study treatment for those with hepatitis B; Active hepatitis C subjects (HCV antibody positive with HCV-RNA levels above the lower limit of detection).

17. Subjects with current active hepatitis B (HBsAg positive with more than 1000 copies /ml(200 IU/ml) of HBV-DNA or higher than the lower limit of detection, whichever is higher) are required to receive anti-HBV therapy during the study treatment for those with hepatitis B; Active hepatitis C subjects (HCV antibody positive with HCV-RNA levels above the lower limit of detection).

18. The history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation is known 19.No remission of toxicity from prior antitumor therapy, defined as toxicity not returning to the level specified in the NCI CTCAE Version 5.0, level 0 or level 1, or in the inclusion/exclusion criteria, except for hair loss in subjects who develop irreversible toxicity and are not expected to be aggravated after administration of the investigational drug (e.g., hearing loss) After consultation, subjects may be included in the study of long-term toxicity caused by radiation therapy, and those who are judged by the investigator to be unable to recover may be included in the study.

20.Known allergy to any component of any investigational drug; There is a known history of severe hypersensitivity to other monoclonal antibodies.

21.If a live or attenuated vaccine has been administered within 30 days prior to the first dose, or if a live or attenuated vaccine is planned to be administered during the study period, inactivated vaccine use is permitted.

22.Known history of mental illness substance abuse alcohol or drugs 23. Pregnant or lactating women 24.The presence of any past or current abnormality in laboratory tests for treatment of disease that may confuse the study results, affect the subject's full participation in the study, or that participation in the study may not be in the subject's best interest.

25.Local or systemic diseases caused by non-malignant tumors; Or disease or symptoms secondary to the tumor that may lead to higher medical risk and/or uncertainty in the evaluation of survival, such as tumor leukemia-like reactions, manifestations of cachexia, etc 26.Any condition that the investigator believes may cause the subject to receive the study drug treatment to be at risk of interfering with the evaluation of the study drug, or affecting the interpretation of the study results。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival assessed by RECIST v1.1 | 6-month
  6-month progression-free survival assessed by RECIST v1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  Objective response rate (ORR)
disease control rate (DCR) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  disease control rate (DCR)
duration of response (DoR) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  duration of response (DoR)
progression-free survival (PFS) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  progression-free survival (PFS)
overall survival (OS) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  overall survival (OS)
Incidence and severity of adverse events (AES) | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  Incidence and severity of adverse events (AES) with clinically significant unusual

OTHER OUTCOMES:
PD-L1 expression | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  PD-L1 expression
MMR status | Until the investigator determines that there is no longer a clinical benefit ， toxicity is intolerable, treatment is completed at 24 months, or other protocol criteria for disco
  MMR status

CONTACTS AND LOCATIONS:
Overall Officials: jingdong zhang, Principal Investigator — China Medical University, China

IPD SHARING:
Plan to Share IPD: No